CLINICAL TRIAL: NCT02265978
Title: CopeSmart: Using Mobile Technology to Promote Positive Mental Health in Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Principal Investigator, Rachel Kenny, PhD Candidate, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GOIPG/2013/450
Record Dates: First submitted 2014-10-07; First posted 2014-10-16 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: General Mental Health and Well-Being
Keywords: Emotional Self-Awareness; Positive Coping; Help-Seeking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CopeSmart (Experimental)
  Interventions: Device: CopeSmart
- Control (No Intervention)

INTERVENTIONS:
Device: CopeSmart — Participants will use the CopeSmart app at least once per day for four weeks
  Arms: CopeSmart

SUMMARY:
This study evaluates the effectiveness of a mental health mobile app (CopeSmart) in promoting positive mental health through emotional self-awareness in adolescents. Participants will be recruited from second-level schools in Ireland. Schools will be randomly assigned to the intervention or control condition. Participants in the intervention condition will use CopeSmart for a four week period. Those in the control condition will not use any mental health app.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 14 and 19 years
* Must be enrolled in second-level education
* Must have access to an iPhone, iTouch or Android mobile device
* Must obtain signed parental consent to participate

Exclusion Criteria:

- No parental consent

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 387 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in levels of emotional self-awareness measured by the Emotional Self-Awareness Scale | Baseline (pre-test), 4 weeks later (post-test) and 8-10 weeks later (follow up)

SECONDARY OUTCOMES:
Changes in frequency of use of positive coping strategies measured by the Coping Strategies Inventory | Baseline (pre-test), 4 weeks later (post-test) and 8-10 weeks later (follow up)
Changes in levels of well-being measured by the WHO-5 Well-Being Index | Baseline (pre-test), 4 weeks later (post-test) and 8-10 weeks later (follow up)
Changes in help-seeking behaviour measured by the General Help-Seeking Questionnaire | Baseline (pre-test), 4 weeks later (post-test) and 8-10 weeks later (follow up)
Changes in levels of emotional distress measured by the Depression, Anxiety and Stress Scale | Baseline (pre-test), 4 weeks later (post-test) and 8-10 weeks later (follow up)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel E Kenny, M.Psych.Sc., Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland

REFERENCES:
- [Derived] Kenny R, Dooley B, Fitzgerald A. Ecological Momentary Assessment of Adolescent Problems, Coping Efficacy, and Mood States Using a Mobile Phone App: An Exploratory Study. JMIR Ment Health. 2016 Nov 29;3(4):e51. doi: 10.2196/mental.6361. PMID 27899340
- See also: Related Info — http://copesmart.com